CLINICAL TRIAL: NCT00791310
Title: Phase 3b,Evaluation of MorphoTEP With the FDG Among Patients in Severe Sepsis of Unspecified Etiology
Brief Title: Evaluation of MorphoTEP With the FDG Among Patients in Severe Sepsis of Unspecified Etiology
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Mr P Boulanger/ Directeur de la Recherche et de l'Innovation, CHU Nancy
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V1 01/03/2008; 2008-A00780-55
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Last update posted 2010-12-31 (Estimated); Status verified 2010-12

CONDITIONS: Severe Sepsis
Keywords: Medical ICU; Severe sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TEP (Experimental): Performance of of TEP coupled to scanner X
  Interventions: Drug: Flucis

INTERVENTIONS:
Drug: Flucis — FDG injected i.v
  Other Names: FDG

SUMMARY:
The objective of this pilot study is to estimate a procedure where the biological samples routinely obtained at the site of suspected infection could be guided by the early realization of a TEP with FDG coupled to scanner X, in patients hospitalized in ICU for severe sepsis of unspecified etiology.

DETAILED DESCRIPTION:
Severe sepsis constitutes the leading cause of mortality in ICU, in particular because a microbial documentation is lacking in about half of the cases.

Tomography by emission of positons, which uses the property of activated macrophages and leucocytes to collect 18F-fluorodeoxyglucose may prove useful to identify the site(s) of infection and then guide sampling.

Thirty patients will be included over 12 months.

Within 24 hours after admission, patients presented with a severe sepsis of still unknown etiology will benefit from the realization of a morphoTEP, including an examination MtOe with the FDG, associated with a conventional scanner X.

Suspected infected sites will then be the subject of sampling when possible. These samples will be send for microbial culture, histology and TREM-1 expression (membrane-bound and soluble form) when appropriate.

The main judgement criteria will be the percentage of the MtOe exams proved to be useful for diagnosis and/or associated with therapeutic modifications.

This pilot study will make it possible to evaluate the interest of the early realization of a TEP/scanner X examination among severe sepsis patients of unknown origin.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized with severe sepsis
* Absence of infected site clearly identified after 48 hours of a conventional diagnosis assessment or suspicion of one or more additional sites
* Indication of scanner X with injection
* Informed consent obtained

Exclusion Criteria:

* Age over 80
* Immunocompromised status
* Surgical intervention within the previous month
* Hemodynamic instability (defined by the use of more than 0.5µg/kg/min vasopressors)
* Severe hypoxia (defined by a PaO2/FiO2 ratio lower than 150)
* Pregnancy
* Patient already included in another protocol
* Anaphylaxis to Flucis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-11; Primary Completion 2010-10 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of TEP exams useful for the diagnosis and/or with therapeutic implications. | 28 days

SECONDARY OUTCOMES:
Percentage of patients for whom local determinations of TREM and sTREM will have made it possible to identify a strong probability of infection of one or more suspected site | 28 days
Reproducibility of the interpretations carried out under the conditions of protocol | 28 days
Frequency of the medical and technical complications associated with the procedure | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: sebastien Gibot, MD, PhD, Principal Investigator — CHU NANCY
Locations (1):
- CHU; Central Hospital, Nancy, France